CLINICAL TRIAL: NCT00520689
Title: Multipurpose Solution Compatibility With a Silicone Hydrogel Lens
Brief Title: Multipurpose Disinfecting Solution Compatibility With a Silicone Hydrogel Contact Lens
Acronym: Amethyst
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Menicon Co., Ltd. (Industry)
Responsible Party: Craig Woods, Research Manager, CCLR
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P/264/07/M
Record Dates: First submitted 2007-08-22; First posted 2007-08-24 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Myopia; Hyperopia
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator)
  Interventions: Device: Silicone Hydrogel Contact Lens
- 2 (Active Comparator)
  Interventions: Device: Silicone Hydrogel Contact Lens
- 3 (Active Comparator)
  Interventions: Device: Silicone Hydrogel Contact Lens
- 4 (Active Comparator)
  Interventions: Device: Silicone Hydrogel Contact Lens

INTERVENTIONS:
Device: Silicone Hydrogel Contact Lens — use of lens over 2 days
  Other Names: Premio

SUMMARY:
The purpose of this study is to verify the compatibility of a silicone hydrogel lens when used with four multipurpose disinfecting solutions (OPTI-FREE® RepleniSH®, ReNu MultiPlus®, Solo-Care Aqua™ and MeniCareTM Soft).

DETAILED DESCRIPTION:
The purpose of this study is to verify the compatibility of a silicone hydrogel lens when used with four multipurpose disinfecting solutions (OPTI-FREE® RepleniSH®, ReNu MultiPlus®, Solo-Care Aqua™ and MeniCareTM Soft) by observing changes within the cornea.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

1. Is at least 17 years old and has full legal capacity to volunteer
2. Has read and signed an information consent letter, after having the opportunity to ask questions and receive acceptable answers
3. Is willing and able to follow instructions and maintain the study appointment schedule
4. Is correctable to a visual acuity of 6/7.5 (20/25) or better (both eyes) with their habitual vision correction
5. Has normal binocular vision (no strabismus, no amblyopia, and anisometropia less than or equal to 1.00 D)
6. Has clear corneas and no active ocular disease
7. Has had an ocular examination in the last two years.
8. Has a functional pair of spectacles
9. Is a current soft lens wearer replacing their lenses at least monthly
10. Has a distance contact lens prescription between +6.00D to -10.00 DS and can be successfully fitted with the study lens
11. Has astigmatism less than or equal to -1.00DC
12. Agrees to wear the study lenses on a daily wear basis

Exclusion Criteria:

A person will be excluded from the study if he/she:

1. Has any signs or symptoms of dry eye
2. Has any clinically significant blepharitis
3. Has undergone corneal refractive surgery
4. Is aphakic
5. Has any systemic disease affecting ocular health
6. Is using any systemic or topical medications that may affect ocular health
7. Is pregnant or lactating
8. Is participating in any other type of clinical or research study
9. Currently wears daily disposable lenses
10. Currently wears lenses on a continuous or extended wear basis
11. Is unable to successfully wear contact lenses without routinely using rewetting drops

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To see if there are any effects on the cornea when using each contact lens/solution combination. | Over 2 days

SECONDARY OUTCOMES:
To quantify comfort and vision ratings with each lens/solution combination. | over 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Fonn, M Optom, Principal Investigator — University of Waterloo; Craig Woods, PhD, Principal Investigator — University of Waterloo
Locations (1):
- Centre for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada